CLINICAL TRIAL: NCT01456858
Title: Insecticide Treated Polyethylene Sheeting for Prevention of Malaria in Emergencies: an Observational Cohort Study in a Refugee Setting in Sierra Leone
Brief Title: Insecticide Treated Polyethylene Sheeting for Prevention of Malaria in Emergencies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Mentor Initiative (Other)
Collaborators: ECHO (Unknown); UNHCR Country Office Freetown (Unknown); World Health Organization (Other); Wageningen University (Other); London School of Hygiene and Tropical Medicine (Other); National Malaria Control Programme Sierra Leone (Unknown); Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TPS_210_202_01033/01034/01035
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2003-11

CONDITIONS: Malaria
Keywords: Malaria Prevention Refugee Emergency; Malaria, Falciparum C03.752.530.650
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Child UPS Largo Camp (Placebo Comparator): Children 4months-36months enrolled who resided in Largo refugee camp under Untreated plastic sheeting (interior wall and ceiling lining)
  Interventions: Other: Untreated Plastic Sheeting
- Child ITPS Largo Camp (Experimental): Children 4months-36months enrolled who resided in Largo refugee camp under Insecticide treated plastic sheeting (interior wall and ceiling lining)
  Interventions: Other: Insecticide Treated Polyethylene Sheeting
- Child UPS Tobanda Camp (Placebo Comparator): Children 4months-36months enrolled who resided in Tobanda refugee camp under Untreated plastic sheeting (ceiling and interior roof lining)
  Interventions: Other: Untreated Plastic Sheeting
- Child ITPS Tobanda Camp (Experimental): Children 4months-36months enrolled who resided in Tobanda refugee camp under Insecticide treated plastic sheeting (ceiling and interior roof lining)
  Interventions: Other: Insecticide Treated Polyethylene Sheeting

INTERVENTIONS:
Other: Insecticide Treated Polyethylene Sheeting — Insecticide Treated Polyethylene Sheeting is based on the standard polyethylene sheeting that is issued routinely as temporary shelter for people affected by emergencies. During manufacture the pyrethroid insecticide, deltamethrin, is extruded with the polyethylene into three-ply laminated sheets, comprising an inner low-density laminate and two, outer high-density laminates. The insecticide release characteristics enable the deltamethrin to diffuse slowly to the outer surfaces and to become available for pick-up by any insect that lands on the surface.
  Other Names: Zerofly
  Arms: Child ITPS Largo Camp; Child ITPS Tobanda Camp
Other: Untreated Plastic Sheeting — Standard polyethylene sheeting that is issued routinely as temporary shelter for people affected by emergencies. Standard untreated plastic sheeting is Identical to ITPS but without the incorporation of insecticide.
  Arms: Child UPS Largo Camp; Child UPS Tobanda Camp

SUMMARY:
A Phase III malaria prevention trial was conducted in two camps of Liberian refugees in Sierra Leone using Insecticide Treated Polyethylene Sheeting (ITPS) or untreated polyethylene sheeting (UPS) randomly deployed to defined sectors of each camp. The ITPS was impregnated with pyrethroid insecticide during manufacture. In Largo camp the ITPS or UPS was attached to inner walls and ceilings of shelters, while in Tobanda the ITPS or UPS was used to line the ceiling and roof only. Cohorts of children up to 3 years of age were cleared of malaria parasites and monitored for up to 8 months post construction for possible malaria re-infection. Installation teams and refugee groups were blinded as to whether the sheeting was insecticide treated or not.

DETAILED DESCRIPTION:
During the last decade public and private sector organisations, under the leadership of the Roll Back Malaria (RBM) Initiative, have recognised the need to work together to bring complementary expertise to the task of identifying and developing vector control tools appropriate to humanitarian crises. Insecticide Treated Polyethylene Sheeting (ITPS), is one such tool emerging from this process and is being produced commercially. ITPS is based on the standard polyethylene sheeting that is issued routinely as temporary shelter for people affected by emergencies. During manufacture the pyrethroid insecticide, deltamethrin, is extruded with the polyethylene into three-ply laminated sheets, comprising an inner low-density laminate and two, outer high-density laminates. The insecticide release characteristics enable the deltamethrin to diffuse slowly to the outer surfaces and to become available for pick-up by any insect that lands on the surface. Consequently ITPS has dual purpose: to provide shelter but with vector-control potential. Deployment and erection of ITPS is done in the same way as standard tarpaulin shelters.

Until now evaluation of ITPS has been limited to small scale entomological testing in scientifically controlled environment 'entomological platforms' in Asian and 'experimental huts' in rural African settings (Refer to Citation Section). Before any novel control tool can go forward for recommendation by the WHO, or be used routinely in humanitarian crises, clear demonstration of impact on malaria morbidity in emergency refugee settings is essential. A Phase III field evaluation was therefore conducted to evaluate the impact of ITPS on malaria incidence in young children in an area of intense transmission. A unique feature of this trial was its setting - a true emergency - in two newly built refugee camps for Liberian refugees displaced to Sierra Leone. The findings offer insight into the effectiveness of ITPS when used in a scenario for which it was purposefully designed.

ELIGIBILITY:
Inclusion Criteria:

* Resident of LARGO or TOBANDA Refugee Camp, Sierra Leone, West Africa
* Child whose guardian has given informed consent for their child to be enrolled into monitoring
* Child aged 4 months to 3 years

Exclusion Criteria:

* Residents who answer "Yes" to the question, "Do you anticipate/plan on moving out of this shelter or camp in the next 6-12 months?"
* Children who have a serious illness other than malaria, based on guardian report.
* Children who have experienced adverse reactions to Amodiaquine or Artesunate on a previous occasion.
* Guardians of children who answer "Yes" to the question, "Do you anticipate/plan on moving out of this shelter or camp in the next 12 months?"

Ages: 4 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2003-12; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Malaria Incidence | 8 months
  The primary outcome was the malaria incidence rate between children in each study arm (ITPS V's UPS) in each refugee camp. Between Dec 2003 and July 2004, daily monitoring of children in both camps was conducted from health screening points. Any child presenting with fever or reported fever in the last 24 hours was administered a clinical questionnaire based on the Integrated Management of Childhood Illness (IMCI), after which a RDT was taken to confirm malaria positivity. Malaria incidence rate was estimated as the total number of malaria episodes per person year over the course of the trial.

SECONDARY OUTCOMES:
Anaemia (From Haemoglobin levels) | 8 months
  In each study cohort (ITPS V's UPS arms in two camps) haemoglobin levels were monitored at 3 monthly intervals (three times during the 8 month monitoring period) using a HemoCue® photometer that was calibrated daily when used.
Adverse Event to ITPS | 8 Months
  Symptoms or conditions considered to be potential adverse events related to ITPS usage (dizziness, inflamed/watery eyes, mucosal irritation, muscle cramps/tremors, nausea, runny nose, skin burning, skin itching, skin paraesthesia, skin rash, skin redness, sneezing and tachycardia (pulse rate >150)) were recorded during the monitoring period in both ITPS and UPS intervention arms in each camp. A symptom listed repeatedly within a seven day period for each child was considered to be the same adverse event as was any child having more than one of the symptoms present on a single day.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Burns, BSc MSc PhD viva pending, Principal Investigator — Wageningen University
Locations (1):
- The Mentor Initiative, Freetown, Sierra Leone

REFERENCES:
- [Result] Graham K, Mohammad N, Rehman H, Nazari A, Ahmad M, Kamal M, Skovmand O, Guillet P, Allan R, Zaim M, Yates A, Lines J, Rowland M. Insecticide-treated plastic tarpaulins for control of malaria vectors in refugee camps. Med Vet Entomol. 2002 Dec;16(4):404-8. doi: 10.1046/j.1365-2915.2002.00395.x. PMID 12510893
- [Result] Diabate A, Chandre F, Rowland M, N'guessan R, Duchon S, Dabire KR, Hougard JM. The indoor use of plastic sheeting pre-impregnated with insecticide for control of malaria vectors. Trop Med Int Health. 2006 May;11(5):597-603. doi: 10.1111/j.1365-3156.2006.01605.x. PMID 16640611
- [Result] Djenontin A, Chabi J, Baldet T, Irish S, Pennetier C, Hougard JM, Corbel V, Akogbeto M, Chandre F. Managing insecticide resistance in malaria vectors by combining carbamate-treated plastic wall sheeting and pyrethroid-treated bed nets. Malar J. 2009 Oct 20;8:233. doi: 10.1186/1475-2875-8-233. PMID 19843332
- [Result] Chandre F, Dabire RK, Hougard JM, Djogbenou LS, Irish SR, Rowland M, N'guessan R. Field efficacy of pyrethroid treated plastic sheeting (durable lining) in combination with long lasting insecticidal nets against malaria vectors. Parasit Vectors. 2010 Aug 3;3(1):65. doi: 10.1186/1756-3305-3-65. PMID 20682050
- [Result] Djenontin A, Chandre F, Dabire KR, Chabi J, N'guessan R, Baldet T, Akogbeto M, Corbel V. Indoor use of plastic sheeting impregnated with carbamate combined with long-lasting insecticidal mosquito nets for the control of pyrethroid-resistant malaria vectors. Am J Trop Med Hyg. 2010 Aug;83(2):266-70. doi: 10.4269/ajtmh.2010.10-0012. PMID 20682865